CLINICAL TRIAL: NCT03476161
Title: A Randomised Controlled Trial Comparing Bond Failure of Buccal Tubes Bonded With Conventional Pre-coated Adhesive vs Flash-free Buccal Tubes
Brief Title: Bond Failure of Two Types of Molar Buccal Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 213576
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): upper left and lower right 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ Flash-Free Adhesive
  upper right and lower left 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ II Adhesive
  Interventions: Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ Flash-Free Adhesive. 4069-6103 / 4069-6114 / 4069-6203 / 4069-6214; Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ II Adhesive. 3069-6103 / 3069-6114 / 3069-6203 / 3069-6214
- Group 2 (Other): upper right and lower left 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ Flash-Free Adhesive
  upper left and lower right 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ II Adhesive
  Interventions: Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ Flash-Free Adhesive. 4069-6103 / 4069-6114 / 4069-6203 / 4069-6214; Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ II Adhesive. 3069-6103 / 3069-6114 / 3069-6203 / 3069-6214

INTERVENTIONS:
Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ Flash-Free Adhesive. 4069-6103 / 4069-6114 / 4069-6203 / 4069-6214 — One type of first permanent molar buccal tube used for fixed orthodontic treatment. One types of adhesive, with same buccal tube base.
Device: 3M Unitek Victory Series™ Superior Fit Buccal Tube with APC™ II Adhesive. 3069-6103 / 3069-6114 / 3069-6203 / 3069-6214 — One type of first permanent molar buccal tube used for fixed orthodontic treatment. One types of adhesive, with same buccal tube base.

SUMMARY:
This study looks at two new types of orthodontic brackets (metal squares of the brace) that have recently been released. Both types have been developed to allow the brackets to stick better to the tooth surface. The difference between the two groups is the adhesive ('glue') that is used. One uses a more conventional type of pre-coated adhesive (APC-II). The other type uses a new flash-free adhesive that does not require the excess to be removed once placed. It is claimed by the manufacturer that this new adhesive has a far lower failure rate than other types. However, there are very few studies that have looked into the bond failures of these adhesives comparatively, with most being lab-based studies outside of the mouth.

The purpose of this study is to investigate which of the two bracket types lasts longest when glued to teeth for brace treatment and if there are any particular reasons why they may fail. This in turn will provide good evidence and research for future use of different bracket types, with an aim to prevent brackets from coming loose as little as possible during treatment. This could potentially result in smoother treatment for the participants and fewer visits.

A total of 56 participants within the Orthodontic Department at Guy's Hospital London, shall be recruited to the trial and randomly placed into one of the two groups. The participants invited to take part in the trial will require fixed braces ('train-tracks') and meet the specific criteria that the investigators are looking for. Once the braces are fitted, regular appointments are made and participants are asked to return for emergency appointments if any of the brace comes loose. The total time for follow-up after the brace is fitted is a maximum of 3 months. The results shall then be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring fixed appliances.
* Patients aged >8 years old

Exclusion Criteria:

* Orthognathic patients requiring bands on first permanent molar teeth.
* Patients with cleft lip/palate or any other craniofacial anomalies.
* Patients already in fixed appliances.
* Patients who have first permanent molars missing.
* Patients with hypoplastic first permanent molars/fluorotic first permanent molars.
* Patients with first permanent molars in crossbite with displacement.
* Patients requiring sectional fixed appliances (not including the molars).
* Patients requiring bands on first permanent molars for TPA, Quadhelix etc.
* Patients who have buccal restorations/crowned first permanent molars.
* Patients who do not speak English fluently or understand written English easily.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in bond failure rate between the two molar buccal tubes. | 3 months
  The primary outcome for this study was to detect failure rates associated with a 3M Unitek APC Flash-free adhesive compared to 3M Unitek APCII adhesive system when bonding first permanent molars with 3M Unitek Victory superior fit buccal tubes.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No